CLINICAL TRIAL: NCT06436885
Title: An Exploratory Study of Efficacy and Safety of Iruplinalkib Tablets in Patients With ROS1 Positive Non-small Cell Lung Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanqiu Zhao, professor of medicine, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-NSCLC-IIT-001
Record Dates: First submitted 2024-05-22; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; ROS1; Iruplinalkib Tablets
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Iruplinaakib tablets should be administered orally at a roughly fixed time each day. Once daily, on an empty stomach or with food, 60mg per dose for days 1 to 7, 180 mg per dose from day 8 if tolerated. Swallow the tablet whole, do not crush, divide or chew the tablet
  Interventions: Drug: Iruplinalkib tablets

INTERVENTIONS:
Drug: Iruplinalkib tablets — Iruplinalkib tablets should be administered orally at a roughly fixed time each day. Once daily, on an empty stomach or with food, 60mg per dose for days 1 to 7, 180 mg per dose from day 8 if tolerated. Swallow the tablet whole, do not crush, divide or chew the tablet
  Other Names: Qi Xin Ke

SUMMARY:
This is a single-arm, open, multicenter exploratory clinical trial to observe and evaluate the efficacy and safety of Iruplinalkib Tablets in patients with ROS1 positive non-small cell lung cancer.

DETAILED DESCRIPTION:
Iruplinalkib Tablets should be administered orally at a roughly fixed time each day. Once daily, on an empty stomach or with food, 60mg per dose for days 1 to 7, 180 mg per dose from day 8 if tolerated. Swallow the tablet whole, do not crush, divide or chew the tablet.

The primary end point was objective response rate

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to join the study and sign the informed consent
2. ≥18 years old
3. Histologically or cytologically confirmed stage III unresectable or stage IV ROS1 positive non-small cell lung cancer
4. The ECOG performance status is 0-2
5. At least one measurable lesion according to RECIST 1.1
6. Can swallow pills normally
7. No brain metastases, or asymptomatic brain metastases, or symptomatic brain metastases that are stable for >4 weeks after treatment
8. The function of vital organs meets the following requirements (no blood component, cell growth factor drugs are allowed within 14 days before the first medication):

   Absolute neutrophil count ≥1.5×109/L Platelet ≥100×109/L Hemoglobin ≥90 g/L Serum albumin ≥30 g/L Serum total bilirubin ≤1.5×ULN ALT and AST≤ 2.5 x ULN; if liver metastasis exists, ALT and AST≤5ULN AKP≤ 2.5×ULN Serum creatinine ≤1.5×ULN International Standardized Ratio (INR) ≤1.5×ULN (not receiving anticoagulation therapy)
9. Non-surgical sterilization or female patients of reproductive age who are required to use a medically approved contraceptive method (such as an IUD, contraceptive pill or condom) during the study treatment period and for 3 months after the end of the study treatment period; Serum or urine HCG tests must be negative for women of childbearing age who have been sterilized without surgery within 7 days prior to the first dose. And must be non-lactation period; For male patients whose partner is a woman of reproductive age, effective contraception should be used during the trial and within 3 months after the last dose of the trial drug

Exclusion Criteria:

1. Patients who are participating in another clinical study or are receiving another investigational drug, or who received the investigational device within 4 weeks prior to the first treatment of our investigational drug. Patients may be included in this study if they are participating in a non-interventional clinical trial
2. Mixed small cell and NSCLC histology
3. Known history or evidence of interstitial lung disease or active non-infectious pneumonia
4. Have had other malignancies within the past 5 years or at the same time (except cured basal cell carcinoma of the skin and cervical carcinoma in situ)
5. Prior surgery or immunotherapy must be completed at least 4 weeks, and radiotherapy must be completed at least 2 weeks before the investigational drug begins
6. Have high blood pressure that is not well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); Allow the above parameters to be achieved through the use of antihypertensive therapy; A history of hypertensive crisis or hypertensive encephalopathy
7. Have clinical symptoms or diseases of heart that are not well controlled, such as: (1) NYHA2 or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, (5) QTc>450ms (male); QTc>470ms (Female)
8. Patients with pleural effusion, ascites, or pericardial effusion requiring drainage can be enrolled if their symptoms are assessed to be stable after drainage
9. Congenital or acquired immune deficiency (such as HIV infection); Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥2000 IU/ml, or hepatitis C virus antibody positive
10. Live vaccine was administered within 4 weeks prior to or possibly during the study period
11. The presence of active gastrointestinal (GI) disease or other conditions that significantly interfere with the absorption, distribution, metabolism, or excretion of the investigational drug
12. Known allergy to the investigational drug or its excipients
13. According to the investigator's judgment, the patient has other factors that may affect the study results or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, and family or social factors, which will affect the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiu Zhao, Study Chair — Henan Cancer Hospital
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China